CLINICAL TRIAL: NCT03464942
Title: A Randomised Phase II Trial Comparing the Efficacy of Single-fraction or Multi-fraction SABR (Stereotactic Ablative Body Radiotherapy) With AteZolizumab in Patients With Advanced Triple nEgative Breast Cancer
Brief Title: Stereotactic Radiation and Immunotherapy in Patients With Advanced Triple Negative Breast Cancer
Acronym: AZTEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/013
Record Dates: First submitted 2018-02-21; First posted 2018-03-14 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Participants with triple negative breast cancer will be randomised to receive either SABR 20Gy in one fraction or 24 Gy in 3 fractions , they will then go onto receive atezolizumab for up to 24 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dose (Active Comparator): SABR 20Gy given as a single dose (to 1 -4 metastases with at least 1 untreated metastasis) followed by atezolizumab (1200 mg) every 3 weeks for 24 months.
  Interventions: Radiation: SABR; Drug: Atezolizumab
- Fractionated Dose (Active Comparator): SABR 24Gy given as 3 fractions (to 1 -4 metastases with at least 1 untreated metastasis) followed by atezolizumab (1200 mg) every 3 weeks for 24 months.
  Interventions: Radiation: SABR; Drug: Atezolizumab

INTERVENTIONS:
Radiation: SABR — Single Dose Group: this group will receive 20 Gy of radiation in a single dose within 10 days of randomisation Fractionated Dose: Participants in this dose will receive a total of 24Gy of radiation given as 3 separate fractions of 8 Gy each.
Drug: Atezolizumab — All participants will commence atezolizumab (within 5 days of last SABR dose) 1200 mg every 3 weeks for 24 months

SUMMARY:
This is a multi-centre, open label, phase 2, randomised controlled trial of patients with advanced triple negative breast cancer (TNBC) who have received no more than one line of chemotherapy (not including neoadjuvant or adjuvant therapy) who will be randomised to be treated with SABR 20Gy in 1# followed by atezolizumab or SABR 24Gy in 3# followed by atezolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a histological or cytological diagnosis of Stage IV TNBC breast cancer (see Appendix 7), defined by ER <1%, PR <1% and HER2 negative on IHC and/or non-amplified by ISH by local lab testing.
2. Written informed consent.
3. Male or female participants aged ≥ 18 years and < 70 years.
4. No more than one prior chemotherapy line in the incurable disease setting. For the purposes of this trial, adjuvant or neoadjuvant chemotherapy does not count as a prior line of therapy but chemotherapy given for residual disease post neoadjuvant chemotherapy is considered as one line.
5. Must be 6 or more months from prior adjuvant, neoadjuvant or post neoadjuvant chemotherapy last dose.
6. At least one measurable lesion as per RECIST 1.1 (see Appendix 1) that is not planned to receive SABR.
7. CT scan (CAP), while body bone scan, and FDG-PET scan evidence of ≥ 2 metastases (with ≥ 1 amenable to SABR).
8. Be willing to provide tissue from a newly obtained core biopsy of a metastatic tumour lesion. Newly-obtained is defined as a specimen obtained up to 60 days prior to randomisation. Patients for whom newly-obtained samples cannot be provided (e.g. inaccessible or patient safety concern) may submit an archived specimen only upon agreement from the CPI).
9. ECOG performance status 0 - 1 (see Appendix 6).
10. Expected life expectancy > 6 months.
11. Female participants of childbearing potential must have a negative urine or serum pregnancy within 7 days of trial randomisation.
12. Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the trial through to 5 months after the last dose of atezolizumab.
13. Male participants must agree to use an adequate method of contraception starting with the first SABR treatment, through to 120 days after the last dose of atezolizumab.
14. Adequate Organ Function as defined in the table below:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
    * Platelets ≥ 100 x 109/L,
    * Hemoglobin* ≥ 90 g/L OR ≥ 9 g/dL (Without transfusion or EPO dependency (within 7 days of assessment),
    * Serum creatinine ≤ 1.5 X ULN OR Measured or calculated Creatinine Clearance** ≥ 60 mL/min if Serum Creatinine >1.5
    * X ULN (Creatinine clearance should be calculated per institutional standard. GFR can also be used in place of creatinine or creatinine clearance - see Attachment 5 - Cockcroft-Gault Formula),
    * Serum Total Bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN if Serum Total Bilirubin > 1.5 ULN

In participants with known Gilbert's syndrome:

* Serum Total Bilirubin ≤ 3.0 X ULN AND Direct Bilirubin ≤ 1.5 X ULN,
* Aspartate Aminotransferase (AST/SGOT) and Alanine Aminotransferase (ALT/SGPT) ≤ 2.5 X ULN OR ≤ 4.0 X ULN if liver metastases are present,
* Albumin > 221 μmol/L OR > 2.5 mg/dL,
* International Normalised Ratio (INR) OR Prothrombin Time (PT) OR Activated Partial Thromboplastin Time (PTT) ≤ 1.5 X
* ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants,
* Lactate dehydrogenase (LDH) ≤2.5 x ULN

Exclusion Criteria:

1. Previous radiotherapy (BED > 30Gy) to an area to be treated.
2. Evidence of active brain metastases. Participants with previously treated brain metastases (with surgical resection, stereotactic radiosurgery or palliative whole brain radiotherapy) may participate, provided they have stable brain metastases defined as 2 imaging studies documenting stability of brain metastasis(es) over > 4 weeks.
3. Intention to treat or requirement for treatment with any chemotherapy agent within ± 3 weeks of trial treatment.

   Note: bisphosphonates or RANKL inhibitors are allowed.
4. Evidence of Spinal Cord Compression.
5. Spinal Instability Neoplastic Score ≥ 7 (see Appendix 4), in a lesion scheduled for SABR treatment unless lesion reviewed by a neurosurgical service and considered stable.
6. Untreated lytic metastases in the neck of the femur that erodes the cortex that is scheduled for SABR treatment.
7. Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent and is planned to receive trial therapy or used an investigational device within 4 weeks of trial treatment
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (> or equal to 10mg prednisolone daily) or any other form of immunosuppressive therapy at time of trial treatment. Note: There must be no intention to commence systemic long-term steroid therapy or any form of immunosuppressive therapy within 7 days prior to the planned first dose of atezolizumab treatment. Note: Single (once off) doses of prophylactic steroid therapy are acceptable.
9. Is planned to receive chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to trial treatment or who has not recovered from adverse events (i.e. AEs not at ≤ Grade 1 or at baseline values) due to a previously administered agent.
10. Has a known additional malignancy that is progressing or requires active treatment.
11. Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).

    Note: Participants with indwelling catheters (e.g., PleurX) are allowed.
12. Has uncontrolled hypercalcemia (> 1.5mmol/L ionized calcium or serum calcium >2.99mmol/L or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab. Note: Participants who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible.
13. Has a significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to Cycle 1, Day 1, unstable arrhythmias or unstable angina. Note: Participants with a known left ventricular ejection fraction (LVEF) < 40% will be excluded.

    Note: Participants with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
14. Has a history of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    Note: Participants with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible Note: Participants with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible Note: Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
    * Rash must cover less than 10% of body surface area (BSA).
    * Disease is well controlled at baseline and only requiring low potency topical steroids.
    * No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids).
15. Has a history of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.

    Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
16. Has an active infection requiring systemic therapy.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through to 5 months after or 120 days after the last dose of trial treatment, for women and men respectively.
20. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
21. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
22. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
23. Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study - Influenza vaccination should be given during influenza season only (example: approximately March to October in the Southern Hemisphere). Participants must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study treatment or within 5 months after the last dose of atezolizumab.
24. Has a known history of active TB (Bacillus Tuberculosis).
25. Known hypersensitivity to atezolizumab or its excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months
  To assess the progression free survival of SABR at a dose of 24Gy in 3# followed by atezolizumab and SABR at a dose of 20Gy in 1# followed by atezolizumab in patients with advanced triple negative breast cancer (TNBC).

SECONDARY OUTCOMES:
Best Objective Response (BOR) between different SABR regimens + atezolizumab | 24 months
  Best objective response (BOR) rate: confirmed complete response (CR) or partial response (PR) as per RECIST 1.1
Incidence of treatment emergent adverse events (safety and tolerability) | 24 months
  Toxicities will be assessed using NCI-CTCAE version 4.03. Tolerability is defined as the time until ceasing treatment due to toxicity.
Progression Free Survival Comparison between different SABR regimens + atezolizumab | 24 Months
  To compare the progression free survival between arms
Duration of Response (DOR) between different SABR regimens + atezolizumab | 24 months
  Duration of response (DoR), defined as time from first occurrence of documented response to disease progression or death in participants who achieve a PR or better as per RECIST 1.1.
Disease Control Rate (DCR) between different SABR regimens + atezolizumab | 24 months
  Disease control (DC), defined as achieving a CR, PR or have had stable disease (SD) for at least 21 weeks prior to any evidence of disease progression, based on RECIST 1.1
Time to Treatment Failure between different SABR regimens + atezolizumab | 24 months
  Time to treatment failure (TTF) defined as the time from randomization until cessation of atezolizumab for any reason including disease progression, treatment toxicity, participant preference or death.
Overall Survival between different SABR regimens + atezolizumab | 24 months
  Overall survival, defined as the time from randomization to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Sherene Loi, Prof, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No